CLINICAL TRIAL: NCT02387424
Title: Phase Two: A Pilot Randomized Trial of Mindfulness-Based Cognitive Therapy for the Prevention of Perinatal Depressive Relapse/Recurrence
Brief Title: Mindfulness-Based Cognitive Therapy for the Prevention of Perinatal Depressive Relapse/Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Emory University (Other); Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sona Dimidjian, Professor and Director, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-0353-02; R34MH083866 (NIH)
Record Dates: First submitted 2015-02-12; First posted 2015-03-13 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Postpartum Depression; Pregnancy; Depression
Keywords: depression; mindfulness; pregnancy; prevention; cognitive behavioral therapy
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBCT-PD (Experimental): Mindfulness-based cognitive therapy adapted for perinatal women (MBCT-PD)
  Interventions: Behavioral: MBCT-PD
- OAR (Active Comparator): Ongoing Assessment and Referral (OAR)
  Interventions: Behavioral: OAR

INTERVENTIONS:
Behavioral: MBCT-PD — The 8-session MBCT protocol, with modifications for use in the context of pregnancy and in anticipation of the postpartum.
  Arms: MBCT-PD
Behavioral: OAR — Ongoing Assessment and Referral (OAR) consists of routine screening and referral to behavioral health services within obstetric clinical settings within Kaiser Permanente (KP) in Colorado and Georgia.
  Arms: OAR

SUMMARY:
Pregnant women with histories of depression are at high risk of depressive relapse/recurrence during the perinatal period, and options for relapse/recurrence prevention are limited. Mindfulness-based cognitive therapy (MBCT) has strong evidence among general populations but has not been studied among at risk pregnant women.

This study is the second phase of a multi-phase project adapting MBCT for perinatal women (MBCT-PD).

DETAILED DESCRIPTION:
Mindfulness-based cognitive therapy (MBCT) represents one of the most important recent developments in the effort to prevent recurrent depression. Explicitly designed to modify core underlying vulnerability factors among recovered individuals with histories of depression, MBCT may have high applicability to the prevention of perinatal depression (PD).

During this phase of the project the investigators will conduct a two-site pilot randomized clinical trial with pregnant women at high-risk of perinatal depression, comparing the efficacy of MBCT-PD to a control group in the prevention of depressive relapse and recurrence. Participants assigned to the control group will receive "ongoing assessment and referral" (OAR), consisting of routine screening and referral to behavioral health services within obstetric clinical settings within Kaiser Permanente (KP) in Colorado and Georgia. The investigators will randomly assign participants at each site to 8 weeks of MBCT-PD or OAR.

During this phase, the investigators will address the following aims:

* Specific Aim 1: To test the primary hypothesis that participants receiving MBCT-PD will experience improved depressive outcomes compared to participants receiving OAR, including lower rates of depressive relapse/recurrence and lower depressive symptom severity as compared to participants receiving OAR.
* Specific Aim 2: To explore the secondary hypotheses that participants receiving MBCT-PD will report improved functioning as compared to participants receiving OAR on a range of secondary outcomes, including indices of anxiety and stress and obstetrical complications.
* Specific Aim 3: To explore potential moderators and mediators of depression outcomes.
* Specific Aim 4: To train and evaluate the ability of behavioral health care providers to administer the MBCT-PD program with fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant up to 32 weeks gestation
* Meeting criteria for prior depression
* Failure to meet criteria for a diagnosis of MDD in the last two months
* Available for group intervention scheduled meetings

Exclusion Criteria:

* Presence of schizophrenia or schizoaffective disorder
* Presence of bipolar disorder or current psychosis
* Presence of organic mental disorder or pervasive developmental delay
* Presence of current eating disorder
* Presence of current substance abuse or dependence
* Presence of antisocial, borderline, or schizotypal personality disorder
* Presence of imminent suicide or homicide risk
* Presence of any other axis I or II disorders that necessitate priority treatment not provided by the study protocol
* Women with any medical conditions that would preclude participation, including high-risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Engagement (class attendance) | Up to 8 weeks
  Engagement is operationalized in-part as class attendance, with completion is defined as attendance at a minimum of four classes, and daily home practice recorded daily as the number of times of practice and type of practice, which are classified as either formal or informal practice.
Client Satisfaction (CSQ-8) | Up to 8 weeks
  Participant satisfaction will be evaluated by the CSQ-8, which is designed to yield a homogeneous estimate of general satisfaction with services. An exit interview also will be completed at 6-months postpartum.
MBCT-PD Adherence Scale (MBCT-PD-AS) | Up to 8 weeks
  Treatment fidelity will be assessed to provide checks on the adequacy of treatment implementation, using the MBCT-PD Adherence Scale.
Change in Depressive Relapse Status: Longitudinal Interval Follow-up Evaluation (LIFE) | Up to 6 months postpartum
  Rate of depressive relapse and time to relapse will be assessed using the LIFE, which provides a retrospective assessment of relapse or recurrence based on a semi-structured interview according to DSM-IV-TR diagnostic criteria.
Change in Edinburgh Postpartum Depression Scale (EPDS) | Up to 6 months postpartum
  Change in the severity of depressive symptoms will be evaluated by the Edinburgh Postpartum Depression Scale (EPDS), which is the most widely used self-report measure of antenatal and postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sona Dimidjian, PhD, Principal Investigator — University of Colorado, Boulder; Sherryl Goodman, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - University of Colorado Boulder, Boulder, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Kaiser Permanente, Atlanta, Georgia